CLINICAL TRIAL: NCT01790191
Title: Comparison of the Effect of Repeated Exposure, Flavor-Flavor Learning and Flavor-Nutrient Learning on Vegetable Acceptance in Weaning Age Infants
Brief Title: Comparison of Effect of Repeated Exposure, Flavor-Flavor and Flavor-Nutrient Learning on Vegetable Acceptance in Infants
Acronym: T221_HabEat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Collaborators: European Union (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: T221_HabEat
Record Dates: First submitted 2013-02-06; First posted 2013-02-13 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Development of Eating Behavior
Keywords: Children; Eating behaviour; Intake; Liking; Conditioned liking; Flavour; Nutrient; Vegetable
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- RE group (Experimental): Repeated consumption of artichoke purée. This group was exposed to basic artichoke puree from Exposure 1 to 10 (E1 to E10)
  Interventions: Behavioral: Repeated consumption of basic artichoke purée.
- FFL group (Active Comparator): Repeated consumption of artichoke purée. This group (Flavor-flavor learning group) was exposed to sweet artichoke puree from Exposure 1 to 10 (E1 to E10).
  Interventions: Behavioral: Repeated consumption of sweet artichoke purée.
- FNL group (Active Comparator): Repeated consumption of artichoke purée. This group (Flavor-nutrient learning group) was exposed to fat, energy-dense artichoke puree from Exposure 1 to 10 (E1 to E10).
  Interventions: Behavioral: Repeated exposure to fat artichoke purée.

INTERVENTIONS:
Behavioral: Repeated consumption of basic artichoke purée. — In this conditioning trial, the effect of repeated consumption of different types of artichoke purée was studied. In Arm 1, participants were repeatedly exposed to basic artichoke purée. In Arm 2, participants were repeatedly exposed to sweet artichoke purée. In Arm 3, participants were repeatedly exposed to fat artichoke purée. Change in intake and liking of basic artichoke purée was evaluated at baseline and after 10 exposures to artichoke purée ; and at 3 follow-ups: after 2 weeks (FU2W), after 3 months (FU3M) and after 6 months (FU6M).
  Arms: RE group
Behavioral: Repeated consumption of sweet artichoke purée. — In this conditioning trial, the effect of repeated consumption of different types of artichoke purée was studied. In Arm 1, participants were repeatedly exposed to basic artichoke purée. In Arm 2, participants were repeatedly exposed to sweet artichoke purée. In Arm 3, participants were repeatedly exposed to fat artichoke purée. Change in intake and liking of basic artichoke purée was evaluated at baseline and after 10 exposures to artichoke purée ; and at 3 follow-ups: after 2 weeks (FU2W), after 3 months (FU3M) and after 6 months (FU6M).
  Arms: FFL group
Behavioral: Repeated exposure to fat artichoke purée. — In this conditioning trial, the effect of repeated consumption of different types of artichoke purée was studied. In Arm 1, participants were repeatedly exposed to basic artichoke purée. In Arm 2, participants were repeatedly exposed to sweet artichoke purée. In Arm 3, participants were repeatedly exposed to fat artichoke purée. Change in intake and liking of basic artichoke purée was evaluated at baseline and after 10 exposures to artichoke purée ; and at 3 follow-ups: after 2 weeks (FU2W), after 3 months (FU3M) and after 6 months (FU6M).
  Arms: FNL group

SUMMARY:
This study aims at comparing learning mechanisms to increase vegetable acceptance in infants at complementary feeding, namely repeated exposure (RE), flavor-flavor learning (FFL) and flavor-nutrient learning (FNL); measuring the stability of the learning effect; and examining the impact of infants' feeding history on vegetable acceptance.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants, aged between 4 and 8 months old, not yet introduced to complementary foods

Exclusion Criteria:

* Infants with food allergies, with chronic health problem, or born before 36 weeks of gestational age

Ages: 4 Months to 8 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2010-10; Primary Completion 2011-07 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Food intake | Participants will be followed for an average duration of 8 months
  Intake of artichoke puree at baseline and at different time points of the experiment (Exposures 1 to 10 defined as E1, E2, E3, E4, E5 ,E6, E7, E8, E9, E10, Postexposure, FU2W, FU3M, FU6M)

SECONDARY OUTCOMES:
Food Liking | Participants will be followed for an average duration of 8 months
  Evolution of Liking of artichoke puree at baseline and at different time points of the experiment (Exposures 1 to 10 defined as E1, E2, E3, E4, E5 ,E6, E7, E8, E9, E10, Postexposure, FU2W, FU3M, FU6M)

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Nicklaus, PhD, Principal Investigator — Centre des Sciences du Goût et de l'Alimentation INRA
Locations (1):
- Centre des Sciences du Goût et de l'Alimentation, Dijon, France

REFERENCES:
- See also: Web site for the main research project funded by the European Union — http://www.habeat.eu/